CLINICAL TRIAL: NCT00061490
Title: The Impact of Weight Loss and Exercise on Knee Osteoarthritis
Brief Title: The Effect of Weight Loss and Exercise on Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: K23AR002160 (NIH); K23AR002160 (NIH); NIAMS-080
Record Dates: First submitted 2003-05-28; First posted 2003-05-29 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Arthritis; Weight Loss
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Arthritis; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 16 weekly educational meetings
  Interventions: Behavioral: Behavioral weight control and lifestyle exercise
- 2 (No Intervention): Wait list control

INTERVENTIONS:
Behavioral: Behavioral weight control and lifestyle exercise — 16 weekly educational meetings vs. waitlist control
  Arms: 1

SUMMARY:
This study will evaluate whether a program of weight loss and exercise can help individuals with knee osteoarthritis (OA).

DETAILED DESCRIPTION:
Knee OA is a major public health challenge affecting millions of people in the United States. Obesity is a primary target for intervention since it accounts for up to 30% of knee OA, exacerbates symptoms, and is associated with bilateral involvement and more rapid progression of the disease. While the American College of Rheumatology (ACR) Practice Guidelines recommend modest weight loss as symptomatic therapy, no published clinical trials have investigated the impact of weight loss on knee OA.

Physical activity has also been associated with pain reduction and increased mobility in individuals with knee OA and the ACR Practice Guidelines indicate that it should be included in treatment. Exercise may be especially helpful for overweight persons with knee OA as it is a potent predictor of weight loss maintenance. Though adherence to traditional exercise programs has been poor, adopting lifestyles in which exercise is accumulated throughout the day appears to be a promising new approach to physical activity. Lifestyle exercise may enhance exercise adherence by increasing options to be active and reducing time barriers. Episodic physical activity may also be preferable to continuous exercise by reducing pain and avoiding injury. The primary objective of this proposal is to evaluate the impact of weight loss and lifestyle exercise on knee osteoarthritis.

Participants will be randomly assigned to either a behavioral weight loss and exercise program or a delayed intervention group. Participants in the behavioral weight loss and exercise group will attend weekly group meetings at the Johns Hopkins Bayview Medical Center for 16 weeks. Group meetings last about 1 hour and are led by health care professionals. Participants will be taught how to lose weight and keep weight off by changing what they eat and evaluating their lifestyle. Participants will be instructed on a safe and effective diet plan (1200 calories/day for women; 1500 calories/day for men) and will be asked to increase their physical activity to about 30 minutes per day of brisk walking, most days of the week. After the 16-week program, groups will continue to meet every three months for 1 year to help sustain lifestyle changes.

The delayed intervention group will receive the program described above after a 4-month waiting period.

The primary outcome measure will be knee pain. Secondary measures include physical disability, quality of life, performance measures, and long-term adherence to behavior change.

ELIGIBILITY:
Inclusion Criteria

* Knee arthritis
* Pain on > 50 % of days in the month in one or both knees
* Difficulty with activities of daily living due to knee pain
* X-ray documenting knee OA within 1 year prior to study entry
* 15 lbs to 50 lbs overweight

Exclusion Criteria

* Significant cardiac, pulmonary, renal, or hepatic disease
* Major psychiatric disease
* ACR functional class IV
* Structured exercise more than once per week for 20 minutes or longer during the 3 months prior to study entry
* Anticipates moving from the area within 18 months of study entry
* Anticipates undergoing knee surgery within 1 year of study entry
* Weight loss of more than 5 kg (11 lbs) in 3 months prior to study entry
* Anorexiant or other medications known to affect metabolism
* Current or planned pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2002-09 (Actual); Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Pain | 4 months and 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan J. Bartlett, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States